CLINICAL TRIAL: NCT02023892
Title: The Effect of Single Dose of Atorvastatin on Change of Circulating Endothelial Microparticles
Brief Title: Single Dose of Atorvastatin and Circulating Endothelial Microparticles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yi-jun Huang, PhD, Department of Pharmacology, Zhongshan School of Medicine, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YHuang002
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Endothelium; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: interventions — Atorvastatin; Sugars; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- atorvastatin (Experimental): atorvastatin 20mg tablet, single dose of 80mg by mouth
  Interventions: Drug: atorvastatin
- placebo (Placebo Comparator): placebo 20mg tablet, single dose of 80mg by mouth
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: atorvastatin
  Other Names: Liptor
  Arms: atorvastatin
Drug: placebo
  Other Names: sugar pill manufactured to mimic atorvastatin 20mg tablet
  Arms: placebo

SUMMARY:
Healthy subjects take single dose of 80mg atorvastatin, then measured their circulating endothelial microparticles and flow-mediated vasodilation in the brachial artery by ultrasound at different time points.

ELIGIBILITY:
Inclusion Criteria:

* healthy youth

Exclusion Criteria:

* acute pathologies
* familial history of cardiovascular disease
* smoking or drinking alcohol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
change of circulating endothelial microparticles | from 1h to 24h after taking atorvastatin